CLINICAL TRIAL: NCT00455962
Title: Effect of Race on Gonadotropin Responses to Short Term Negative and Positive Feedback Effects of Gonadal Steroids
Brief Title: Effect of Race on Gonadotropin Responses
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Clinical Associate in Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2003P-001397; Sundry Department Fund (Other: MGH-REU Department Fund); R01AG013241 (NIH)
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Premenopause; Healthy
Keywords: estrogen; progesterone; African-American; Caucasian; infusion; gonadotropins; healthy

STUDY DESIGN:
Intervention Model Description: Comparisons will be made between response to estradiol and progesterone infusion in young African-American and Caucasian women.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- African American women 18-35 yo (Active Comparator): intervention: estradiol steroid infusion and progesterone steroid infusion
  Interventions: Drug: Estradiol steroid infusion; Drug: Progesterone steroid infusion
- Caucasian women 18-35 yo (Active Comparator): intervention: estradiol steroid infusion intervention: progesterone steroid infusion
  Interventions: Drug: Estradiol steroid infusion; Drug: Progesterone steroid infusion

INTERVENTIONS:
Drug: Estradiol steroid infusion — Estradiol infusion of 0.1 mcg/kg/hr for 12 hr, 0.135 mcg/kg/hr for 12 hr, 0.165 mcg/kg/hr for 12 hr and 0.2 mcg/kg/hr for 60 hr
  Other Names: E2
Drug: Progesterone steroid infusion — Progesterone infusion of 4.77 nmol/kg/hr (1.5 mcg/kg/hr) for 24 hr and 6.36 nmol/kg/hr (2 mcg/kg/hr) for the final 24 hr
  Other Names: P

SUMMARY:
The purpose of this study is to attempt to determine why estrogen levels are increased in African-American women as compared to Caucasian women by evaluating estrogen feedback on the brain. African-American women have increased bone mineral density, higher rates of twins, greater incidence of fibroids, and increased incidence of breast cancer below 40 years of age as compared to Caucasian women. These traits or illnesses are all believed to be estrogen-dependent. In fact, previous research has demonstrated increased estrogen levels in African-American women as compared to Caucasian women. However, the reason for these differences in estrogen levels has not been studied in humans. One possibility is that estrogen feedback on the brain differs between African-American and Caucasian women. Two small glands in the brain (hypothalamus and pituitary) respond to estrogen. The hypothalamus secretes GnRH (Gonadotropin-Releasing Hormone) that signals the pituitary to secrete the reproductive hormones, LH (Luteinizing Hormone) and FSH (Follicle Stimulating Hormone). These hormones act on the ovaries and signal the ovaries to produce estrogen and progesterone. Estrogen in the bloodstream then acts on the brain to stop this system when the blood has enough estrogen levels. This is called estrogen feedback. This study will determine whether there are differences in estrogen feedback between African-American and Caucasian women.

DETAILED DESCRIPTION:
Several independent lines of evidence have suggested that reproductive endocrine dynamics may differ between African-American (AAW) and Caucasian (CW) women. There is an increased incidence of dizygotic twinning in African-American women and a further increase in the incidence reported in African women compared to Caucasian, Hispanic and Asian populations. While the etiology of dizygotic twinning is not well understood, an increase in its incidence may imply an alteration in the integrated control of the reproductive axis which usually favors development of a single ovulatory follicle. It is widely appreciated that the incidence of leiomyomas is increased in African-American women. Growth factors are likely to play a role in their control, but there is also ample evidence that leiomyomas are responsive to gonadal steroids, decreasing in size following the menopause and in response to hypoestrogenism caused by gonadotropin downregulation. African-American women under 40 years of age have a higher risk of breast cancer than women of all other ethnicities in that age group, again raising the question of whether there are also differences in reproductive hormone dynamics. Finally, bone density is increased in African-American women. In a cross-sectional study of 54 African-American and 39 Caucasian women between the ages of 20 and 90, Perry et al found that the increase in bone density in AAW was associated with increased serum levels of both estradiol and testosterone. Woods et al also described increased levels of estradiol, estrone and androstenedione levels in AAW compared with control women on a controlled low-fat, high-fiber diet. In contrast, a recent longitudinal cohort study has suggested that AAW have lower levels of estradiol with increasing age and BMI in comparison with CW. We have compared reproductive hormone levels in AAW and CW < 35 years old with a history of regular ovulatory cycles. Our preliminary data indicate that in comparison to age and BMI matched CW, estradiol levels are consistently elevated across the cycle in AAW in the absence of changes in LH, FSH, progesterone, inhibin A or inhibin B. These relationships suggest both altered negative and forward feedback interrelationships between FSH and LH and estradiol in the setting of normal inhibin levels. In the current protocol we will seek to understand the mechanisms underlying these feedback differences, which have never been addressed in these populations.

A graded infusion of estradiol and progesterone can be used to assess differences in negative and positive feedback of gonadal steroids on LH and FSH. We have hypothesized that differences exist in feedback regulation of the hypothalamus and pituitary as a function of African-American or Caucasian race in reproductive aged women.

ELIGIBILITY:
Inclusion Criteria:

* African-American women aged 18 to 35 years and Caucasian women aged 18 to 36 years. Subjects will be asked to volunteer information on ethnicity (self classification). Only African-American and Caucasian subjects will be included in this aim to address the specific hypotheses.
* BMI <30
* In good general health with normal TSH, prolactin and hemoglobin
* Normal BUN and Creatinine (< 2 times the upper limit of normal)
* On no medications for > 2 months before the study
* Regular menstrual cycles every 25 to 35 days and ovulation documented by a luteal phase progesterone > 3 ng/ml
* Willing to use abstinence or barrier methods of contraception for the duration of the study.

Exclusion criteria:

* postmenopausal
* smoking >9 cigarettes per day
* evidence of androgen excess.
* sensitivity to any medications used in the relevant protocol
* race other than African-American or Caucasian
* Hispanic ethnicity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 23 (Actual)
Dates: Start 2005-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Coded individual level data with all identifiers removed will be available on request to the PI.

REFERENCES:
- [Result] Shaw ND, Klingman KM, Srouji SS, Histed SN, Hall JE. Gonadotropin responses to estrogen-positive and -negative feedback are identical in African-American and Caucasian women. J Clin Endocrinol Metab. 2012 Jan;97(1):E106-9. doi: 10.1210/jc.2011-2102. Epub 2011 Nov 2. PMID 22049179

RESULTS

PARTICIPANT FLOW:
Groups:
- African American Women: Healthy African-American women 18-35 years old
  Estradiol steroid infusion: Estradiol infusion of 0.1 mcg/kg/hr for 12 hr, 0.135 mcg/kg/hr for 12 hr, 0.165 mcg/kg/hr for 12 hr and 0.2 mcg/kg/hr for 60 hr
  Progesterone steroid infusion: Progesterone infusion of 4.77 nmol/kg/hr (1.5 mcg/kg/hr) for 24 hr and 6.36 nmol/kg/hr (2 mcg/kg/hr) for the final 24 hr
- Caucasian Women: Healthy Caucasian women 18-35 years old
  Estradiol steroid infusion: Estradiol infusion of 0.1 mcg/kg/hr for 12 hr, 0.135 mcg/kg/hr for 12 hr, 0.165 mcg/kg/hr for 12 hr and 0.2 mcg/kg/hr for 60 hr
  Progesterone steroid infusion: Progesterone infusion of 4.77 nmol/kg/hr (1.5 mcg/kg/hr) for 24 hr and 6.36 nmol/kg/hr (2 mcg/kg/hr) for the final 24 hr
Period: Overall Study
Arm/Group | African American Women | Caucasian Women
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African American Women | Caucasian Women | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Continuous [Mean (Full Range); unit: years] | 28 [22 to 36] | 28 [23 to 36] | 28 [22 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 0 | 10
  White | 0 | 13 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: LH Peak in Response to Estrogen Positive Feedback
Description: Estradiol levels are consistently higher in African-American vs Caucasian women across the menstrual cycle. This study was designed to determine if African-American women are more sensitive to estrogen positive feedback to generate the preovulatory LH surge using a controlled estrogen infusion paradigm.
Time Frame: 5 days of estradiol and progesterone infusion
Population: Healthy African-American and Caucasian women aged 18-35 with regular ovulatory menstrual cycles.
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | African American Women | Caucasian Women
Number analyzed (Participants) | 10 | 13
IU/L | 80.3 (13.3) | 73.1 (11.6)
Statistical Analysis 1: Comparison: African American Women vs Caucasian Women; Using previously collected data from a group of 18 predominantly Caucasian women undergoing a similar infusion we determined that 22 women would be necessary to identify a 30% difference in peak LH levels, the primary outcome measure, between AAW and CW with 80% power at a significance level of 0.05; Test type: Superiority; p = 0.69, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | African American Women | Caucasian Women
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No